CLINICAL TRIAL: NCT03576677
Title: Effect of Levosimendan or Placebo on Exercise Capacity and Hemodynamics in Patients With Advanced Chronic Heart Failure (LOCO-CHF Trial)
Brief Title: Effect of Levosimendan or Placebo on Exercise in Advanced Chronic Heart Failure
Acronym: LOCO-CHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Finn Gustafsson (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor-Investigator, Finn Gustafsson, MD, PhD, DMSci, Professor of Cardiology, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RH-HJE-LN-02
Record Dates: First submitted 2018-06-11; First posted 2018-07-03 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
Keywords: Advanced chronic heart failure; Exercise capacity; Exercise hemodynamics; Levosimendan
MeSH Terms: conditions — Heart Failure | interventions — Simendan

STUDY DESIGN:
Intervention Model Description: This is a prospective multi-center, double-blinded, placebo controlled, randomized study in patients with advanced chronic heart failure. Patients who meet the eligibility criteria will be randomized in a 1:1 ratio for treatment with 6 hours infusion of either (i) levosimendan 0.2 µg/kg/min or (ii) placebo (sterile 5% dextrose).
  At baseline an upright ergometer maximal exercise test is performed to determine max workload and pVO2 (Test 0). Based on this test 50% of pVO2 with corresponding workload (watt) is calculated (submax).
  At Day 0 patients will perform a supine ergometer maximal exercise test (Test 1) with simultaneous invasive hemodynamic measurement by Swan-Ganz catheter. Subsequently, patients will receive 6 hours infusion of study medication.
  At Day 5 (4-6 days after infusion of study medication) patients will repeat the supine ergometer maximal exercise test (Test 2) with simultaneous invasive hemodynamic measurements.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blinded; hence neither patients nor investigators are aware of the treatment assignment throughout the study period. 2 unblinded study nurses at each site will perform randomization and prepare study medication blinded to the rest of the research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levosimendan (Active Comparator): Study participants in this arm will receive a 6 hours infusion of levosimendan 0.2 µg/kg/min.
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): Study participants in this arm will receive a 6 hours infusion of placebo (sterile isotonic sodium chloride + 5% dextrose + vitamin B)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan — Levosimendan, 2.5 mg/mL concentrate for dilution. 5 mL of the study drug will be injected into a 245 mL isotonic glucose solution.
  Patients will receive a 6 hours infusion of this study drug at an infusion rate of 0.2 µg/kg/min.
  Other Names: Simdax
  Arms: Levosimendan
Drug: Placebo — The placebo solution will be prepared by adding 10 mL of 5% dextrose to a vial containing Soluvit (vitamin B) under aseptical conditions. 5 mL of this solution is then added to 245 mL of isotonic sodium chloride solution.
  5% dextrose and vitamin B are added to ensure yellow coloring indistinguishable from the active drug (levosimendan).
  Patients will receive a 6 hours infusion of this study drug. Infusion rate will be calculated in similar fashion to the levosimendan group.
  Arms: Placebo

SUMMARY:
Purpose: This study evaluates the subacute effect of levosimendan infusion on exercise capacity and exercise hemodynamics compared with placebo in patients with advanced chronic heart failure.

Hypothesis: Treatment with 6 hours infusion of levosimendan compared with placebo improves exercise capacity and exercise hemodynamics evaluated by change in CO/PCWP.

Design: The study is a prospective multi-center, double-blinded, placebo controlled randomized study. 42 consecutive patients who meet the eligibility criteria will be enrolled.

DETAILED DESCRIPTION:
Background: Patients with advanced heart failure (HF) symptoms (NYHA III-IV) have poor quality of life and significantly impaired functional capacity despite optimal medical management. Exercise intolerance in HF results from multiple pathophysiological processes, but central hemodynamics during exercise are important determinants. In patients with advanced HF, intermittent levosimendan infusion is sometimes used to relieve symptoms and possibly improve prognosis. A short-term effect of levosimendan infusion on exercise capacity has previously been reported. However, the underlying mechanisms behind such an improvement, as well as more durable effects of levosimendan on exercise capacity in advanced chronic HF, have not been clearly established. Also the hemodynamic effect of levosimendan has not been investigated in advanced chronic HF during exercise.

To our knowledge no previous studies have evaluated the subacute effect of levosimendan infusion on exercise capacity and exercise hemodynamics in patients with advanced chronic HF. This study will hopefully improve the understanding of the role of levosimendan in the management of these patients.

Purpose: This study evaluates the subacute effect of levosimendan infusion on exercise capacity and exercise hemodynamics compared with placebo in patients with advanced chronic HF.

Hypothesis: Treatment with 6 hours infusion of levosimendan 0.2 µg/kg/min compared with placebo improves exercise capacity and exercise hemodynamics evaluated by change in CO/PCWP (Day 0 to Day 5 (4-6) after infusion) in patients with advanced chronic HF.

Design: The study is a prospective multi-center, double-blinded, placebo controlled randomized study. The study population will consist of 42 consecutive patients who meet the eligibility criteria. Patients will be randomized 1:1 to treatment with either levosimendan or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* NYHA III-IV on optimal medical treatment
* LVEF ≤35%
* NT-proBNP >600 µg/L
* pVO2 <20 mL/kg/min
* No hospitalization for HF or change in loop diuretic <2 weeks

Exclusion Criteria:

* Recent or acute coronary and respiratory syndromes
* Recent sustained ventricular tachycardia or ventricular fibrillation
* Severe aortic or mitral valve disease
* Known malfunctioning artificial heart valve
* Uncorrected obstructive valvular disease
* Hypertrophic cardiomyopathy
* Fertile women
* Uncorrected thyroid disease
* Presence of any disease/condition that might per se influence exercise performance
* Left ventricular assist device
* Pacemaker-guided heart rate at rest or during exercise
* Known contraindication for treatment with levosimendan
* Any treatment with levosimendan in the previous 6 months
* Inability to perform a VO2max test
* Symptomatic hypotension or systolic blood pressure < 90 mmHg

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
ΔCO/PCWP (submax) | Day 0 to Day 5 (4-6)
  Change in CO/PCWP from Day 0 (infusion of study medication) to Day 5 (day 4-6) at the workload corresponding to 50% of pVO2 determined at baseline

SECONDARY OUTCOMES:
ΔCO/PCWP (peak) | Day 0 to Day 5 (4-6)
  Change in CO/PCWP from Day 0 (infusion of study medication) to Day 5 (day 4-6) at peak exercise
ΔCO (peak) | Day 0 to Day 5 (4-6)
  Change in maximal CO from Day 0 (infusion of study medication) to Day 5 (day 4-6) at peak exercise
ΔPCWP (peak) | Day 0 to Day 5 (4-6)
  Change in PCWP from Day 0 (infusion of study medication) to Day 5 (day 4-6) at the maximal load obtained during both invasive measurements
CO maximal | Day 5
  Maximal CO at Day 5 (day 4-6)
PCWP maximal | Day 5
  Maximal PCWP at Day 5 (day 4-6)
SvO2 maximal | Day 5
  Maximal SvO2 at Day 5 (day 4-6)
Workload maximal | Day 5
  Maximal workload (watt) at Day 5 (day 4-6)
ΔPCWP (rest) | Day 0 to Day 5 (4-6)
  Change in resting PCWP from Day 0 (infusion of study medication) to Day 5 (day 4-6)
ΔCO (rest) | Day 0 to Day 5 (4-6)
  Change in resting CO from Day 0 (infusion of study medication) to Day 5 (day 4-6)
ΔCVP (rest) | Day 0 to Day 5 (4-6)
  Change in resting CVP from Day 0 (infusion of study medication) to Day 5 (day 4-6)
ΔmPA (rest) | Day 0 to Day 5 (4-6)
  Change in resting mPA from Day 0 (infusion of study medication) to Day 5 (day 4-6)
ΔSvO2 (rest) | Day 0 to Day 5 (4-6)
  Change in resting SvO2 from Day 0 (infusion of study medication) to Day 5 (day 4-6)
Δ6MWT day 3 | Day 0 to Day 3
  Change in 6MWT from Day 0 (infusion of study medication) to Day 3
Δ6MWT day 5 (4-6) | Day 0 to Day 5 (day 4-6)
  Change in 6MWT from Day 0 (infusion of study medication) to Day 5 (day 4-6)
Δ6MWT day 14 | Day 0 to Day 14
  Change in 6MWT from Day 0 (infusion of study medication) to Day 14
ΔNT-proBNP day 3 | Day 0 to Day 3
  Change in NT-proBNP from Day 0 (infusion of study medication) to Day 3
ΔNT-proBNP day 5 | Day 0 to Day 5 (day 4-6)
  Change in NT-proBNP from Day 0 (infusion of study medication) to Day 5 (day 4-6)
ΔNT-proBNP day 14 | Day 0 to Day 14
  Change in NT-proBNP from Day 0 (infusion of study medication) to Day 14
QOL day 3 | Day 3
  Quality of life (QOL) score using the Kansas City Cardiomyopathy Questionnaire (KCCQ) at Day 3 after infusion of study medication
QOL day 5 | Day 5
  Quality of life (QOL) score using the Kansas City Cardiomyopathy Questionnaire (KCCQ) at Day 5 (4-6) after infusion of study medication
QOL Day 14 | Day 14
  Quality of life (QOL) score using the Kansas City Cardiomyopathy Questionnaire (KCCQ) at Day 14 after infusion of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD, professor, PhD, DMSci, Principal Investigator — Department of Cardiology, The Heart Center, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark
Locations (3):
- Denmark (3):
  - Department of Cardiology, The Heart Center, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Department of Cardiology, Copenhagen University Hospital, Herlev and Gentofte Hospital, Herlev, Denmark, Herlev
  - Department of Cardiology, Odense University Hospital, Odense, Denmark, Odense